CLINICAL TRIAL: NCT02715999
Title: Transversus Abdominis Plane Versus Quadratus Lumborum Block for Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Gözen Öksüz, Associate Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 05-02/2016
Record Dates: First submitted 2016-03-13; First posted 2016-03-22 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quadratus Lumborum Block (Active Comparator): Quadratus Lumborum block group (QL) patients will receive unilaterally Quadratus Lumborum block using Bupivacaine 0.2 %
  Interventions: Procedure: Quadratus Lumborum Block
- Transversus abdominis plane block (Active Comparator): Transversus abdominis plane block (TAP) patients will receive unilaterally TAP block using Bupivacaine 0.2 %
  Interventions: Procedure: Transversus Abdominis Plane Block

INTERVENTIONS:
Procedure: Quadratus Lumborum Block — After preoxygenation for three minutes, anesthesia would be induced with 8% sevoflurane inhalation in 50% oxygen and % 50 air ; 1ug/kg fentanyl and 3 mg/kg propofol is administered intravenously. Then laryngeal mask is inserted when conditions are satisfactory.All patients will be in the lateral position . Under ultrasound guidance a 22 Gauge, Pajunk Sonoplex(medical Germany) needle will be used for both techniques. Under ultrasound 0.5 ml/kg bupivacaine 0.2 % injected unilaterally at the posterior border of the quadratus lumborum muscle
  Other Names: QLB
  Arms: Quadratus Lumborum Block
Procedure: Transversus Abdominis Plane Block — After preoxygenation for three minutes, anesthesia would be induced with 8% sevoflurane inhalation in 50% oxygen and % 50 air ; 1ug/kg fentanyl and 3 mg/kg propofol is administered intravenously. Then laryngeal mask is inserted when conditions are satisfactory. All patients will be in the lateral position . Under ultrasound guidance a 22 Gauge, Pajunk Sonoplex(medical Germany) needle will be used for both techniques. Under ultrasound 0.5 ml/kg bupivacaine 0.2 % injected unilaterally between internal oblique and transversus abdominis muscles.
  Other Names: TAP
  Arms: Transversus abdominis plane block

SUMMARY:
The purpose of this research study is to find the best way to decrease pain in children whom have had low abdominal surgery. Investigators will perform two technique of trunk block; Transversus abdominis plane or Quadratus lumborum block .The method used is often chosen by which one the doctor has more experience using. The Investigator plans to find out if one of the methods is more effective and/or safer than the other method.

The results of this study will help learn how to best control pain in children having surgery low abdominal surgery.

DETAILED DESCRIPTION:
Children aged 1-7 years undergoing lower abdominal surgeries would be recruited in this randomized study.

Children would be monitored by electrocardiogram, pulse oximeter and non-invasive blood pressure.

After preoxygenation for three minutes, anesthesia would be induced with 8% sevoflurane inhalation in 50% oxygen and % 50 air ; 1ug/kg fentanyl and 3 mg/kg propofol is administered intravenously. Then laryngeal mask is inserted when conditions are satisfactory (jaw relaxed, lash reflex disappeared, no coughing, gagging, swallowing).After ethical committee approval, informed written consent will be obtained from all patients.

Consenting patients scheduled to have unilaterally low abdominal surgery(inguinal hernia,hydrocele,undescended testicles surgery will be randomised to unilateral Quadratus lumborum block or Transversus abdominis plane block at the begin of surgery.

All patients will be in the lateral position . Under ultrasound guidance a 22 Gauge, Pajunk Sonoplex(medical Germany) needle will be used for both techniques. The spread of injectate will be seed on ultrasound.The dose of local anaesthetic in both groups will be 0.5 ml/kg 0.2 % Bupivacaine. Anesthesia would be maintained with 2% sevoflurane An increase in blood pressure or heart rate by more than 15% from preoperative value was defined as insufficient analgesia and was treated with fentanyl 0.5 µ/kg. Saline dextrose 5% (1:1) solution was infused in a dose of 12 ml/ kg /h.

All patients heart rate,MAP and Oxygen saturation record intraoperatively. All patients will receive paracetamol if requirement for postoperative analgesia.All patient will transfer from PACU to day-surgery unit (DSU) if they achieved Modified Aldrete Score of ten.

All patients will be assessed postoperatively by a blinded investigator: in the postanesthesia care unit and at 30 min 1,2, 4, 6, 12, 24, hour postoperatively.FLACC score will be used.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* undergoing unilateral low abdominal surgery

Exclusion Criteria:

* history of allergic reactions to local anesthetics
* rash or infection at the injection site
* anatomical abnormality
* bleeding diatheses, coagulopathy, liver diseases

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
time to first use of analgesic | 24 hour
  By investigators until hospital discharge, then through telephone interview with parents after that

SECONDARY OUTCOMES:
Total paracetamol consumption | 24 hour
  By investigators until hospital discharge, then through telephone interview with parents after that
Parent satisfaction scores | 24 hour
  By investigators until hospital discharge, then through telephone interview with parents after that
FLACC (face, legs, activity, cry, consolability) | 1,2,4,6,12,24 hour
  By investigators until hospital discharge, then through telephone interview with parents after that

CONTACTS AND LOCATIONS:
Overall Officials: Gözen Öksüz, M.D., Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University Hospital, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Derived] Oksuz G, Bilal B, Gurkan Y, Urfalioglu A, Arslan M, Gisi G, Oksuz H. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block in Children Undergoing Low Abdominal Surgery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):674-679. doi: 10.1097/AAP.0000000000000645. PMID 28759502